CLINICAL TRIAL: NCT01794494
Title: Prospective Observation Study of Patient Outcome and Cost Effectiveness of Interventions for Critical Ischemia
Brief Title: Prospective Observation Study of Outcome of Interventions for Critical Ischemia
Acronym: PROVENCE
Status: Completed | Type: Observational
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Klas Osterberg, Dr, Sahlgrenska University Hospital
Other Study IDs: PROVENCE-1
Record Dates: First submitted 2013-02-09; First posted 2013-02-20 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Critical Limb Ischemia
Keywords: Peripheal arterial disease; Critical limb ischemia; Bypass surgery; Subintimal angioplasty; Health related cost
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia | interventions — Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Open surgical group: Bypass surgery for critical limb ischemia
  Interventions: Procedure: Bypass surgery
- Endovascular treatment: Endovascular recanalization for critical limb ischemia
  Interventions: Procedure: Endovascular recanalization

INTERVENTIONS:
Procedure: Bypass surgery — Patients are treated with femoro-popliteal bypass
  Groups: Open surgical group
Procedure: Endovascular recanalization — Patients are treated with PTA or subintimal angioplasty
  Groups: Endovascular treatment

SUMMARY:
Severe atherosclerosis in the leg arteries is termed critical limb ischemia (CLI). This condition gives great suffering for the patients in terms of pain, wounds and often developing gangrene. Untreated, the condition has a high risk of amputation. In Sweden, the majority of the patients are investigated and evaluated for treatment. Treatment is carried out either by traditional open bypass surgery or balloon dilatation technology (endovascular treatment). The latter method is still under development, and studies have shown that the treatment has less local and systemic complications than bypass surgery. It is also shown that the method has a limitation in that the treatment effect is less durable. What is the role of minimally invasive technologies should have in the future is unclear, mainly due to its efficiency and cost-effectiveness compared with bypass surgery are not evaluated. In a prospective observational study we intend study the effectiveness, cost-effectiveness and impact on quality of life in patients undergoing treatment for critical CLI with bypass surgery or endovascular treatment in Västra Götaland Region (VGR). All patients over a period of two years, which undergo treatment for CLI with either of the two methods will be included in the study. Patients will be followed up with regard to the clinical efficacy and health-related quality of life after treatment at, respectively one, 12 and 24 and 60 months. Cumulative care costs are calculated and estimates of cost are made. This study aims to increase knowledge about the role of endovascular treatment of CLI shall have in the future.

DETAILED DESCRIPTION:
Prospective Observation Study of Cost Effectiveness of Interventions for Critical Ischemia

Background The incidence of arteriosclerotic disease increases with age and is one of society's greatest public health problem. Impaired circulation to the lower limbs, termed peripheral arterial disease (PAD) is a common diagnosis in the older populations. Estimates show that about 10% of the population over age 70 suffers from symptomatic PAD. [1] Milder forms of the disease causes walking induced pain in the legs, termed intermittent claudication, resulting in a variable restriction of walking ability. As the disease progresses, circulatory impairment becoming more pronounced, often resulting in rest pain, impaired wound healing, or in the worst cases gangrene. These latter stages of PAD categorized as critical limb ischemia, is usually followed by a pronounced reduction in the individual's mobility and quality of life. The incidence of critical limb ischemia in Sweden is estimated at about 40 per 100 000 inhabitants, which means that each year more than 600 individuals in the Västra Götaland Region (VGR) suffer from this condition. [2] Untreated critical ischemia leads to a high risk of amputations. Investigations of the blood circulation of these patients arterial circulation generally reveal extensive arteriosclerotic vascular lesions including arterial occlusions (stop) in the vessels supplying the lower extremities. Interventions designed to improve blood flow has ability to reduce symptoms and in the short or long term eliminate amputation threat. The established treatment principle has since the 1960s been bypass surgery. The method involves major open surgery, including a period of hospitalization and has a high incidence of local as well as general complications.

Since more than a decade, a minimally invasive technique to restore flow in occluded artery has become widely used. The method termed as subintimal angioplasty (SAP) uses catheter and guide wire to get through the occluded vessel section, followed by balloon dilatation. The method is under development and increases in use both internationally and in Sweden. The advantage is that the procedure has less risk for local and systemic complications. The procedures is also associated with shorter hospital stays. Disadvantages are that the duration of treatment is often shorter and the procedure often has to be repeated. [3] It is currently unknown if Endovascular intervention is a cost effective way to treat critical limb ischemia. Furthermore, the impact on patient health-related quality of life (HRQL) is in the short and long term unknown. What role the minimally invasive technologies will have in the future is unclear, mainly due to that efficiency and cost-effectiveness compared to bypass surgery have not thoroughly been evaluated, which was pointed out in a national health technology assessment "Benartärsjukdom - diagnosis and treatment". [1]

Purpose The purpose of this study is to evaluate the effectiveness, cost efficiency, and patient benefits including HRQL in the short and long term for the two principally different methods of treatment for critical limb ischemia in as far as possible unselected clinical population of VGR. The effectiveness of treatment methods are evaluated for their ability to prevent amputations, provide symptom improvement, duration of treatment (patency), cumulative health care cost up to two years, and the effects on HRQL.

Question / Hypothesis

1. Endovascular treatment for CLI is comparable with open bypass surgery for limb salvage
2. Endovascular treatment for CLI is comparable with open bypass surgery for alleviating CLI symptoms
3. Endovascular treatment is associated with better HRQL in the short term and comparable HRQL in the long term (two years) compared with open bypass surgery.
4. Endovascular treatment of CLI is a cost-effective option as compared to open bypass surgery

A clinical study of structure as below can identify selection criteria for the method to be offered to the patient as the primary method for critical limb

Method: Sample / Representativeness The survey is conducted in the form of a prospective observational study in which the two cohorts followed for two years.

Inclusion criteria: patients with CLI due to arterial occlusion of the superficial femoral artery and popliteal artery being considered for bypass surgery or SAP at any of the four vascular surgical units in VGR.

Exclusion criteria: Patients with occlusions at levels above the origin of the superficial femoral artery or occlusions, which has a distribution more distal to the popliteal artery. Patients with inability to understand patient information for informed consent.

A prospective randomized study with high internal validity, are often considered to have greater value than a controlled comparative observational study. The problem is that the external validity tends to be low in prospective randomized trials often only a small percentage of patients can be randomized between the two treatments.

The difficulties of a prospective randomized study on this type of question can be exemplified by the BASIL study where only 20% of patients requiring treatment for CLI were randomized into the study. [4] The advantage of a prospective observational study is that substantially all of the patients in the region being treated for critical limb ischemia and that do not satisfy the exclusion criteria can be included, so that the external validity is high, and that the results may be implemented in the clinical practice.

Inclusion of patients is made on the four units over two years, in connection with decisions on treatment. In total 250 patients under 2 years will be included in the study.

Method: Grouping The analysis divided subjects into those who bypass surgery and those who have undergone endovascular treatment.

Methods: The intervention Bypass Surgery: The operation is an open surgical procedure that is performed under general anesthesia or regional anesthesia. [5] This method means that the blood is bypassed the occluded artery by a new vessel (usually vein).

Angioplasty: Using intra arterial catheter technology, a guide wire and catheter is passed through the occluded vessel section. Balloon dilatation will thereafter recreate a new channel for blood flow. [6] The surgery is a minimally invasive procedure that is done under local anesthesia.

Method: Data Collection Initial data collection: General information as age, presence of diabetes, hypertension, heart disease, and smoking obtained.

A validated scale, the Rutherford scale together with ankle pressure, assesses the degree of CLI. [7] Anatomic mapping of the vessel lesions before revascularization is performed by digital subtraction angiography, MRI or CT scan.

In order to rate the extent of the arterial lesions the preoperative investigations were examined with respect to

* starting point of occlusion
* length of the occlusion
* the distal arterial run-off (number of open leg vessels). These data form the basis for subsequent matching of populations.

Prospective follow-up:

Clinical Evaluation: The two treatment groups had followed up at one, 12, 24 and 60 months. At these time points, patients were examined with ankle pressure, ultrasound (duplex) and clinical condition (possibly amputation, ischemic degree of Rutherford scale). Any additional treatment for arterial occlusion or to prevent occlusion of during the study period was registered.

The costs of treatment are followed prospectively in the Regional Health Database. After follow-up, a calculation of treatment costs for each patient. Health-related quality of life: data obtained before treatment, after 1 month and after 24 months using Vascular Quality of Life Questionnaire (VascuQol) that is designed for use in peripheral arterial disease and EQ 5D.

Method: Data Processing

The treatment effect is estimated in the two groups with respect to:

* amputation free survival
* patency
* clinical symptoms
* cumulative health care cost and QALY for the two different treatment options
* HRQoL

Clinical follow-up in accordance with the DEFINE group consensus document for follow-up after treatment of lower limb ischemia. [7] After statistical matching of the population on the basis of the prospective data variables, a comparative analysis is performed. Special analysis is made of the patient population in which both methods are deemed to have been possible to implement.

Cumulative cost of care: Both the costs and effects of both the methods will be studied. Costs will be followed in the Regional Health Database for admissions related to the two interventions. The cost of complications will be assigned patients under gross-costing method, which means that the price per action and cost per complication will be the same for all patients. In other words, it is therefore only the number and type of measure and number and type of complication that will affect the cost of each treatment arm. This does not affect the outcome of patient-specific factors that are not related to the question in the study. Efficacy will be based on measurements using the EQ-5D and the result of the measurement can be transformed into utilities which in turn can be used to calculate quality-adjusted life years (QALYs). [8, 9] Health-related quality of life: VascuQol is designed for use in peripheral arterial disease including CLI. The questionnaire consists of 25 questions in 5 domains (pain, symptoms, activities, social and emotional). [11]

Expected Results / Significance Critical ischemia is a common cause of pain, ulceration and gangrene of the lower extremities in the elderly. The disease causes great suffering for the victims and leads to large social costs in the form of high hospitalization consumption.

For patients with CLI, treatment with bypass surgery has been the standard treatment for decades. The results are suboptimal, data from Swedish vascular register, Swedvasc shows that 3% die within a month, 18% are not improved, 10% are amputees within a year. Over the past 10-15 years, the technique of endovascular treatment, known as subintimal angioplasty, developed and spread to more and more clinics. The method is increasingly being used as first-line treatment of critical limb ischemia, despite lack evidence of its efficiency and cost effectiveness. As healthcare resources are limited, it is essential that a new treatment is evaluated before it is introduced as a routine method. For ethical reasons and resource reasons, it is essential that patients with severe disease may receive, in both the short and long term, the most effective treatment. This study aims to clarify the effectiveness of both bypass surgery and endovascular treatment of critical limb ischemia due to occlusion of the superficial femoral artery and / or knee artery in a clinical normal population.

ELIGIBILITY:
Inclusion Criteria:

* patients with CLI due to arterial occlusion of the superficial femoral artery and/or the popliteal artery being considered for bypass surgery or SAP at any of the four vascular surgical units in VGR.

Exclusion Criteria:

* patients with CLI due to arterial occlusion of the aorto-iliac arterial segment or distal to the politeal segment.
* Patients with inability to understand patientinformation and informed concens.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with critical limb ischemia coming to the for vascular department in the western region of Sweden.
Sampling Method: Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Amputation-free survival | 2 years
  Freedom of death and amputation during the study

SECONDARY OUTCOMES:
Change in Rutherford scale | 2 Years
  Change in Rutherford scale from baseline:International established scoring system 0-6 for grading of lower limb ischemia.

OTHER OUTCOMES:
Rate of re-intervention | 2 years
  Primary patency: Freedom from occlusion of bypass-graft or endovacular treated arterial segment and freedom of restenosis that need intervention in bypass-graft or endovascular treated arterial segment.
  Secondary patency:Freedom from occlusion of bypass-graft or endovacular treated arterial segment. Treated for restenosis in bypass-graft or endovascular treated arterial segment.
Health related quality of life | 2 years
  Health related quality of life measured by VASCUQOL. VascuQol consists of 25 items, subdivided into five domains. Each question has a seven-point response scale. The responses are averaged to give an overall and a domain score ranging from one (worst Health Related Quality of Life, HRQoL) to seven (best HRQoL).
Health related quality of life | 2 years
  Health related quality of life measured by EQ-5D-3L. EuroQol- 5 dimensions (EQ-5D-3L) consists of 5 items, subdivided into five domains. Each question has a three-point response scale. The score is used to calculate an index between 0 (worst HR) to 1 (best HRQoL).
Cost effectiveness | 2 years
  Cumulative health care costs in dollars

CONTACTS AND LOCATIONS:
Overall Officials: Klas Österberg, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Department of vascular surgery, Sahlgrenska University Hospital, Gothenborg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1.Benartärsjukdom diagnostics and treatment. A systematic literature review. 2007: SBU. Swedish Council on Technology Assessment.
- [Background] Barani J, Mattiasson I, Lindblad B, Gottsater A. Suboptimal treatment of risk factor for atherosclerosis in critical limb ischemia. Int Angiol. 2005 Mar;24(1):59-63. PMID 15877000
- [Background] Met R, Van Lienden KP, Koelemay MJ, Bipat S, Legemate DA, Reekers JA. Subintimal angioplasty for peripheral arterial occlusive disease: a systematic review. Cardiovasc Intervent Radiol. 2008 Jul-Aug;31(4):687-97. doi: 10.1007/s00270-008-9331-7. Epub 2008 Apr 15. PMID 18414946
- [Background] Adam DJ, Beard JD, Cleveland T, Bell J, Bradbury AW, Forbes JF, Fowkes FG, Gillepsie I, Ruckley CV, Raab G, Storkey H; BASIL trial participants. Bypass versus angioplasty in severe ischaemia of the leg (BASIL): multicentre, randomised controlled trial. Lancet. 2005 Dec 3;366(9501):1925-34. doi: 10.1016/S0140-6736(05)67704-5. PMID 16325694
- [Background] KUNLIN J. [Long vein transplantation in treatment of ischemia caused by arteritis]. Rev Chir. 1951 Jul-Aug;70(7-8):206-35. No abstract available. Undetermined Language. PMID 14865345
- [Background] Bolia A, Miles KA, Brennan J, Bell PR. Percutaneous transluminal angioplasty of occlusions of the femoral and popliteal arteries by subintimal dissection. Cardiovasc Intervent Radiol. 1990 Dec;13(6):357-63. doi: 10.1007/BF02578675. PMID 2149672
- [Background] Diehm N, Pattynama PM, Jaff MR, Cremonesi A, Becker GJ, Hopkins LN, Mahler F, Talen A, Cardella JF, Ramee S, van Sambeek M, Vermassen F, Biamino G. Clinical endpoints in peripheral endovascular revascularization trials: a case for standardized definitions. Eur J Vasc Endovasc Surg. 2008 Oct;36(4):409-19. doi: 10.1016/j.ejvs.2008.06.020. Epub 2008 Aug 8. PMID 18692415
- [Background] Bjoholt I, Janson M, Jonsson B, Haglind E. Principles for the design of the economic evaluation of COLOR II: an international clinical trial in surgery comparing laparoscopic and open surgery in rectal cancer. Int J Technol Assess Health Care. 2006 Winter;22(1):130-5. doi: 10.1017/s0266462306050926. PMID 16673689
- [Background] Sullivan M, KJTC, SF-36 Health Survey: Manual and Interpretation Swedish Guide, Second Edition, Göteborg: Sahlgrenska University Hospital
- [Background] Morgan MB, Crayford T, Murrin B, Fraser SC. Developing the Vascular Quality of Life Questionnaire: a new disease-specific quality of life measure for use in lower limb ischemia. J Vasc Surg. 2001 Apr;33(4):679-87. doi: 10.1067/mva.2001.112326. PMID 11296317